CLINICAL TRIAL: NCT02780908
Title: Cardio-respiratory Responses During Hypoxic Exercise in Individuals Born Prematurely
Acronym: PreTerm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jozef Stefan Institute (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other); University Medical Centre Ljubljana (Other); University of Lausanne (Other); University of Lyon (Other); Lancaster University (Other); University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JozefSI
Record Dates: First submitted 2016-05-19; First posted 2016-05-24 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Hypoxia; Altitude Sickness; Tolerance
MeSH Terms: conditions — Hypoxia; Altitude Sickness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypoxia at rest and exercise (Experimental): The participants will perform a resting test, hypoxia sensitivity test and a graded exercise test to voluntary exhaustion in normoxic condition ((HYPO; FiO2=0.120 corresponding to terrestrial altitude of approx. 4000 m)
  Interventions: Other: Graded exercise testing; Other: Resting testing
- Normoxia at rest and exercise (Placebo Comparator): The participants will perform a resting test and a graded exercise test to voluntary exhaustion in normoxic condition ((NORM; fraction of inspired oxygen (FiO2)=0.209, placebo)
  Interventions: Other: Graded exercise testing; Other: Resting testing

INTERVENTIONS:
Other: Graded exercise testing — All graded exercise tests will be performed on electromagnetically controlled cycle-ergometer Ergo Bike Premium. The testing protocol will commence with a 10-min resting period, to obtain the resting cardio-respiratory values, followed by a 5-min warm up at a work rate of 60 W. Thereafter the workload will increase every fourth minute by 40 W. The participants will be required to maintain a cadence of 60·min-1 throughout the whole test. The test is terminated when the participant is unable to maintain the assigned cadence.
Other: Resting testing — The resting test will be performed in supine position with participants breathing normoxic air (FiO2=0.21) for 30 min and hypoxic gas for the subsequent 30-min (FiO2=0.120). During the whole protocol duration the respiration, local blood flow, ECG and EEG will be measured non-invasively.

SUMMARY:
This project will consist of two studies, each investigating resting and exercise cardio-respiratory responses during exposure to hypoxia in individuals born prematurely and individuals born at full term of two different age groups: Kids (10-14 yrs) and Adults (18-22 yrs).Additional study will be performed on a preterm adult cohort (15 participants) that will investigate potential differences between hypobaric and normobaric hypoxia as outlined in the following section.

DETAILED DESCRIPTION:
The study protocol in each age group will comprise two visits to the laboratory testing sessions in a randomized order. On one occasion the participants will perform a resting hypoxia test and a graded exercise test to voluntary exhaustion in normoxic condition ((NORM; fraction of inspired oxygen (FiO2)=0.209, placebo). On a second visit the participants will perform a hypoxia sensitivity test and a graded exercise test to voluntary exhaustion in hypoxic condition (HYPO; FiO2=0.120 corresponding to terrestrial altitude of approx. 4000 m). Indirect calorimetry, near infrared spectroscopy and ECG measurements will be performed throughout all tests. During both testing sessions the participants will also undergo anthropometry measurements and pulmonary function testing. The outline of the research visits is presented in the bellow figure:

ELIGIBILITY:
Inclusion Criteria:

Healthy male individuals

PRETERM group; gestational age: ≤ 32 weeks; gestational weight ≤ 1500 g

CONTROL group: full term born individuals ≤ 38 weeks

Exclusion Criteria:

Medication required that may interfere with the interpretation of the results

Chronically illnesses

Hormonal therapy

Recent sub-standard nutritional status

Family history of respiratiory, cardio-vascular, renal or hematological disease History of: thyroid dysfunction, renal stones, diabetes, allergies, hypertension, hypocalcaemia, uric acidaemia, lipidaemia or hyperhomocystinaemia

History of mental illness

Smoker within six months prior to the start of the study

Abuse of drugs, medicine or alcohol

Participation in another study up to two months before study onset

No signed consent form before the onset of the experiment

Blood donors in the past three months before the onset of the experiment

Vegetarian and Vegans

Migraines

History of vestibular disorders

Claustrophobia

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Tolerance to hypoxia during rest and exercise in preterm and full term individuals | Two year
  All graded exercise tests will be performed on electromagnetically controlled cycle-ergometer Ergo Bike Premium.The participants will be required to maintain a cadence of 60·min-1 throughout the whole test. The test is terminated when the participant is unable to maintain the assigned cadence. The resting test will be performed in supine position with participants breathing normoxic air (FiO2=0.21) for 30 min and hypoxic gas for the subsequent 30-min (FiO2=0.120). During the whole protocol duration the respiration, local blood flow, ECG and EEG will be measured non-invasively. The resting test will be performed in supine position with participants breathing normoxic air (FiO2=0.21) for 30 min and hypoxic gas for the subsequent 30-min (FiO2=0.120). During the whole protocol duration the respiration, local blood flow, ECG and EEG will be measured non-invasively.
Cardio-respiratory control at rest in normoxia and hypoxia in preterm and full term individuals | One year
  The resting test will be performed in supine position with participants breathing normoxic air (FiO2=0.21) for 30 min and hypoxic gas for the subsequent 30-min (FiO2=0.120). During the whole protocol duration the respiration, local blood flow, ECG and EEG will be measured non-invasively. The resting test will be performed in supine position with participants breathing normoxic air (FiO2=0.21) for 30 min and hypoxic gas for the subsequent 30-min (FiO2=0.120). During the whole protocol duration the respiration, local blood flow, ECG and EEG will be measured non-invasively.

SECONDARY OUTCOMES:
Oxidative stress responses to hypoxic exercise in preterm and full term | One year
  Blood sampling will be performed during each visit at four time points (before and after each test, as detailed on the bellow figure. Besides general hematological markers (CBC, ferritin, transferrin etc.) oxidative stress (advanced oxidation protein products, malondialdehyde and nitrotyrosine) and antioxidant system markers (superoxide dismutase, catalase, ferric-reducing antioxidant power, glutathione peroxidase and uric acid) will be determined as described previously (3). Select gene polymorphisms and their association with the above mentioned oxidative stress markers will also be assessed from the collected blood samples in collaboration with the laboratory for Pharmacogenetics, Medical Faculty, UL
Sensitivity to hypoxia during rest and exercise - Richalet test | One year
  This test will assess individuals tolerance to hypoxia and HVR. As noted in the above figure the test consist of a 4-min periods of normoxic (FiO2=0.210) and hypoxic (FiO2=0.120) rest and hypoxic and normoxic low-intensity exercise. Respiration, gas exchange and capillary oxygen saturation will be measured during the course of the test.
Changes in intestinal metabolites as a result of hypoxic exposure | One year
  The aim of this protocol is to assess whether there are significant differences in physiological status of intestinal metabolites (reducing sugars, short chain fatty acids, amino-acids, index of molecular weight, polyphenols, sterols) between the two populations in response to normoxic and hypoxic testing procedures. As sampling needs to be conducted during the period preceding the actual days of experiments and after the completion of testing, i.e. during the daily routines of participants, auto-sampling protocol was selected as the only option through which samples of feces and urine are going to be collected by participants three days before and after physical testing.
Differences between normobaric and hypobaric hypoxia in preterm individuals | Two years
  This part of the study will investigate potential differences between normobaric and hypobaric exposure to hypoxia in preterm born individuals. For this purpose the participants will perform another laboratory visit in Ljubljana and will also be exposed to hypobaric hypoxia in a physiology lab at Aiguille du Midi, which is run by our collaborators. As noted in the bellow schematic each exposure will last 8-hours and measures of respiration, gas exchange and blood sampling will be performed at 2-4 hour periods during the exposure. The participants will be transferred to Chamonix using a van with our research team in groups of four. The transfer from Chamonix to Aiguille du Midi laboratory will be performed via cable car

CONTACTS AND LOCATIONS:
Overall Officials: Damjan Osredkar, MD, PhD, Principal Investigator — University Children's Hospital Ljubljana Department of Pediatric Neurology
Locations (2):
- Slovenia (2):
  - Jozef Stefan Institute, Ljubljana, Ljubljana
  - University Children's Hospital Ljubljana Department of Pediatric Neurology, Ljubljana, Ljubljana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Debevec T, Pialoux V, Mekjavic IB, Eiken O, Mury P, Millet GP. Moderate exercise blunts oxidative stress induced by normobaric hypoxic confinement. Med Sci Sports Exerc. 2014 Jan;46(1):33-41. doi: 10.1249/MSS.0b013e31829f87ef. PMID 23846158
- [Background] Debevec T, Mekjavic IB. Short intermittent hypoxic exposures augment ventilation but do not alter regional cerebral and muscle oxygenation during hypoxic exercise. Respir Physiol Neurobiol. 2012 Apr 30;181(2):132-42. doi: 10.1016/j.resp.2012.02.008. Epub 2012 Mar 2. PMID 22406250
- [Background] Debevec T, Keramidas ME, Norman B, Gustafsson T, Eiken O, Mekjavic IB. Acute short-term hyperoxia followed by mild hypoxia does not increase EPO production: resolving the "normobaric oxygen paradox". Eur J Appl Physiol. 2012 Mar;112(3):1059-65. doi: 10.1007/s00421-011-2060-7. Epub 2011 Jul 7. PMID 21735214
- [Background] Debevec T, Amon M, Keramidas ME, Kounalakis SN, Pisot R, Mekjavic IB. Normoxic and hypoxic performance following 4 weeks of normobaric hypoxic training. Aviat Space Environ Med. 2010 Apr;81(4):387-93. doi: 10.3357/asem.2660.2010. PMID 20377142
- [Background] Debevec T, Pialoux V, Ehrstrom S, Ribon A, Eiken O, Mekjavic IB, Millet GP. FemHab: The effects of bed rest and hypoxia on oxidative stress in healthy women. J Appl Physiol (1985). 2016 Apr 15;120(8):930-8. doi: 10.1152/japplphysiol.00919.2015. Epub 2016 Jan 21. PMID 26796757
- [Background] Debevec T, Simpson EJ, Macdonald IA, Eiken O, Mekjavic IB. Exercise training during normobaric hypoxic confinement does not alter hormonal appetite regulation. PLoS One. 2014 Jun 2;9(6):e98874. doi: 10.1371/journal.pone.0098874. eCollection 2014. PMID 24887106
- [Background] Osredkar D, Sabir H, Falck M, Wood T, Maes E, Flatebo T, Puchades M, Thoresen M. Hypothermia Does Not Reverse Cellular Responses Caused by Lipopolysaccharide in Neonatal Hypoxic-Ischaemic Brain Injury. Dev Neurosci. 2015;37(4-5):390-7. doi: 10.1159/000430860. Epub 2015 Jun 12. PMID 26087775
- [Background] Osredkar D, Thoresen M, Maes E, Flatebo T, Elstad M, Sabir H. Hypothermia is not neuroprotective after infection-sensitized neonatal hypoxic-ischemic brain injury. Resuscitation. 2014 Apr;85(4):567-72. doi: 10.1016/j.resuscitation.2013.12.006. Epub 2013 Dec 19. PMID 24361672
- [Derived] Debevec T, Pialoux V, Poussel M, Willis SJ, Martin A, Osredkar D, Millet GP. Cardio-respiratory, oxidative stress and acute mountain sickness responses to normobaric and hypobaric hypoxia in prematurely born adults. Eur J Appl Physiol. 2020 Jun;120(6):1341-1355. doi: 10.1007/s00421-020-04366-w. Epub 2020 Apr 8. PMID 32270264